CLINICAL TRIAL: NCT02222103
Title: Pilot Study of the MultiSense Patch to Record Cardiopulmonary Data During Sleep and Wake Cycles
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Scripps Clinic (Other)
Responsible Party: Principal Investigator, Steven Steinhubl, Director, Digital Medicine, Scripps Translational Science Institute
Other Study IDs: RDS-Sleep Apnea
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected obstructive sleep apnea in adults: Already scheduled in-lab sleep study

SUMMARY:
The investigators are proposing to use a wearable device, MultiSenseTM, developed by Rhythm Diagnostic Systems, Inc. which has many sensors inside in a "Band-Aid" like strip in order to see if it can help diagnose capabilities in individuals suspected of having obstructive sleep apnea. The MultiSenseTM sensor is a self-contained, reusable, rechargeable, battery-powered, flexible strip, measuring 4 X 1.2 inches that simultaneously tracks and records a number of physiological health related parameters such as ECG, heart rate, pulse synchronized oxygen saturation, temperature, respiratory rate, depth of respiration and motion/position. One advantage of this device over current home diagnostic systems is the capability for recording over several nights.

The objective is to compare multiple biometric parameters tracked by the MultiSenseTM to gold standard monitoring in an accredited sleep lab using polysomnography. Home monitoring will explore potential findings supportive of sleep apnea while monitoring at home during routine sleep over 5 to 7 nights. Enrolling 10 adults already scheduled for a medically indicated sleep study will help us to make these determinations. Subjects will wear the device, which is the size of a Band-Aid, via adhesive to their chest over a period of 10 days. Subjects will go about their normal daily activities and return the device via mail once completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Considered to be at high likelihood for sleep apnea and already scheduled for a formal sleep study.

Exclusion Criteria:

* Congestive heart failure or other major medical illness that would complicate the diagnosis of OSA.
* Psychological or social situation that would make the study difficult for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be adults men and women suspected of having obstructive sleep apnea and already scheduled for an in-lab sleep study at the Scripps Clinic Viterbi Family Sleep Center.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Direct Comparison of MultiSenseTM to Polysomnography for detection of sleep apnea | 10 days
  To compare multiple biometric parameters tracked by the MultiSenseTM to gold-standard monitoring in an accredited sleep lab using polysomnography.

SECONDARY OUTCOMES:
Home monitoring | 10 days
  Explore potential findings supportive of sleep apnea while monitoring at home during routine sleep over 5 to 7 nights.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinhubl, MD, Principal Investigator — STSI
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States